CLINICAL TRIAL: NCT06180694
Title: Reminiscence Therapy Applied to Individuals With Dementia
Brief Title: Reminiscence Therapy in Individuals With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: amasyau-mçy-001
Record Dates: First submitted 2023-12-13; First posted 2023-12-22 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reminiscence group (Experimental): Reminiscence therapies will be applied to individuals with dementia
  Interventions: Other: Reminiscence therapy

INTERVENTIONS:
Other: Reminiscence therapy — Reminiscence therapies will be applied to individuals with dementia in 45-minute sessions once a week for 8 weeks.

SUMMARY:
This research will be carried out with the aim of determining the effect of reminiscence therapy applied to individuals with dementia on cognitive functions, anxiety, depression and activities of daily living.

The research will be conducted with a pre-test post-test single group, quasi-experimental research design.

DETAILED DESCRIPTION:
Dementia; It is a disease that requires intensive use of health services, has a high care burden, and has medical, social, psychological and economic burdens for the patient, family and society. Dementia is characterized by many disorders in cognitive functions, especially memory, thought and social skills. Progressive disorders in cognitive functions cause behavioral changes, decrease in activities of daily living, and neuropsychiatric symptoms such as anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with mild to moderate dementia according to DSM-5 criteria (whether individuals have an official diagnosis of neurocognitive disorder according to DSM-5 criteria and their medical diagnosis will be verified from the health records at the institution),
* Getting a score between 13-23 for the educated (literate) and 10-23 for the uneducated (illiterate) on the mini mental state examination,
* Being 65 years of age or older,
* Being able to communicate,
* No vision or hearing problems,
* Consent to participate in the research.

Exclusion Criteria:

* Getting a score below 13 and above 23 for the educated (literate) and below 10 and above 23 for the uneducated (illiterate) from the mini mental state examination,
* Having an acute illness that prevents participation in intervention sessions,
* Having serious sensory and physical limitations that prevent participation,
* Having severe neuropsychiatric symptoms (agitation, psychosis, apathy, uncontrolled delirium, etc.),
* Having a traumatic life history,
* Having recently participated in a similar program.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Cognitive Status on the Standardized Mini Mental Test (SMMT) at Week 8 | Baseline and week 8
  SMMT, which allows assessing cognitive status, is the most frequently used and easily applied test in dementia screening. The scale is evaluated out of 30 points in total. For SMMT, scores of 23/24 are considered the cutoff score for dementia, but traditionally scores between 24 and 30 are considered normal. A score below 24 indicates cognitive impairment, between 18 and 23 points is considered mild dementia, between 13 and 17 points is considered moderate dementia, and below 12 points is considered severe dementia. Change = (Week 8 Score-Baseline Score)
Change from Baseline in Anxiety Symptoms on Geriatric Anxiety Scale (GAS) | Baseline and week 8
  GAS,developed for the elderly, is a 30-item scale that has somatic, cognitive and affective subscales and monitors anxiety symptoms. The total score on the scale varies between 0-75. A high score indicates a high level of anxiety.Change = (Week 8 Score-Baseline Score)
Change from Baseline in Depressive Symptoms on Geriatric Depression Scale Short Form (GDS-SF) | Baseline and week 8
  GDS-SF, is a scale consisting of 15 questions that questions the emotional state of elderly individuals. The cut-off point of the scale is 7 points and above. Scores between 0 and 4 indicate no depressive symptoms, scores between 5 and 8 indicate mild depressive symptoms, scores between 9 and 11 indicate moderate depressive symptoms, and scores of 12 and above indicate severe depressive symptoms. Change = (Week 8 Score-Baseline Score)
Change from Baseline in Patient's Dependency on Basic Self-Care Behaviors on Katz's Activities of Daily Living Index (KADLI) | Baseline and week 8
  KADLI, evaluates the patient's dependence on basic self-care behaviors that are required to live and are expected to do every day. The scale evaluates the degree of dependency in basic daily living activity parameters, including information on bathing, dressing, toileting, transfer, continence and nutrition. Scoring of the index ranges from 0 to 6, and a patient with a score of 6 is considered independent, and a patient with a score of 0 is considered fully dependent. Change = (Week 8 Score-Baseline Score)

CONTACTS AND LOCATIONS:
Overall Officials: Merve çayır yılmaz, asst. prof., Principal Investigator — Amasya University
Locations (1):
- Merve Çayır Yılmaz, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No